CLINICAL TRIAL: NCT00786435
Title: Carbohydrate Metabolism Impairments in Chronic Human Spinal Cord Injury
Brief Title: Carbohydrate Study, Chronic SCI
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Kim Anderson, Assistant Adjunct Professor, University of California, Irvine
Other Study IDs: 2006-5395
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Those with a cervical spinal cord injury
- 2: Those with a thoracic spinal cord injury
- 3: Healthy, control group

SUMMARY:
As people with spinal cord injuries (SCI) get older they become more likely to develop health problems, just like everyone else. However, SCI increases the risk of certain problems. This research project will focus on the control of blood sugar after SCI. Sugar in the blood is the important source of energy for the body. Too much sugar in the blood is known as hyperglycemia and not enough sugar in the blood is known as hypoglycemia. Under healthy conditions, the amount of sugar in the blood is automatically regulated so that a steady level is maintained. After SCI, however, this automatic regulation is damaged. The likelihood of experiencing too much or too little blood sugar is increased. Over time, having too much blood sugar can lead to the development of diabetes. In just the opposite situation, individuals with SCI can begin to experience more frequent episodes of too little blood sugar. It is thought that the level of SCI, amount of time post-injury, and amount of body fat are important factors in the development of hyperglycemia or hypoglycemia. This study will test 2 of those factors, level of SCI and amount of body fat. A total of 35 subjects will be enrolled, 24 with SCI and 11 able-bodied controls. All procedures will be performed at the university's clinical research center. Susceptibility to hyperglycemia will be tested by having each subject drink a sugar water solution and then taking blood samples every 30 minutes for 2 hours. Hypoglycemia will be tested by very carefully inducing low blood sugar, taking blood samples over a 2 hour time period to evaluate different chemicals, and answering a questionnaire about different symptoms experienced during the procedure. Body fat will be measured by having a special kind of x-ray. It is predicted that subjects with cervical injuries and with more body fat will be at the greatest risk of experiencing hyperglycemia and hypoglycemia. The results from this study will provide important information for future studies aimed at examining the effect of exercise and other potentially therapeutic agents on blood sugar regulation in the aging SCI population.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 5 or more years post-injury.
2. Must have a C1-C8 or T7-T12/L1 lesion.
3. Must be ASIA Impairment Scale grade A or B.
4. Must not require the use of a ventilator.
5. Must not have type I or II diabetes.
6. Must not have any current pressure sores.
7. Must be cognitively competent and have no concomitant brain damage.
8. The study physician will determine for each subject whether any medications will preclude her/him from study participation. Any subject taking anti-cholinergic medication will be asked to not take that medication after midnight prior to study day 2 (they can take it following the hypoglycemia challenge on study day 2).

Exclusion Criteria:

1. Fetuses.
2. Neonates.
3. Pregnant women; a negative pregnancy test will be required for all potential female subjects in reproductive years.
4. Prisoners.
5. Cognitively impaired adults.
6. Institutionalized individuals.
7. Children under age 18.
8. Non-English speaking individuals.
9. Anyone taking lipid altering medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The characteristics of the proposed subject population are that all subjects must be 18-65 years old, male or female, pass a medical examination by the study physician, and must speak English.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2007-08; Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Irvine, California, United States